CLINICAL TRIAL: NCT02884544
Title: Phase II, Open-label, Dose-titration, Safety Study Designed to Determine the Evening Dose of a Novel Delayed and Extended Release Formulation of Dextroamphetamine Sulfate (HLD100) to Produce Optimal Clinical Effects in Children With ADHD
Brief Title: A Study of Delayed and Extended Release Formulation of Dextroamphetamine Sulfate (HLD100) in Children With ADHD
Acronym: HLD100-103
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironshore Pharmaceuticals and Development, Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLD100-103
Record Dates: First submitted 2016-07-28; First posted 2016-08-31 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Attention-Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dextroamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HLD100 10mg (Experimental): HLD100 (dextroamphetamine sulfate) DR/ER capsules (10mg)
  Interventions: Drug: HLD100
- HLD100 20mg (Experimental): HLD100 (dextroamphetamine sulfate) DR/ER capsules (20mg)
  Interventions: Drug: HLD100
- HLD100 30mg (Experimental): HLD100 (dextroamphetamine sulfate) DR/ER capsules (30mg)
  Interventions: Drug: HLD100
- HLD100 40mg (Experimental): HLD100 (dextroamphetamine sulfate) DR/ER capsules (40mg)
  Interventions: Drug: HLD100

INTERVENTIONS:
Drug: HLD100 — Treatment
  Other Names: Dextroamphetamine sulfate, delayed release/extended release

SUMMARY:
The phase 2 study will evaluate the safety, tolerability and efficacy of HLD100 at steady state (following up to 5 weeks of treatment) in children using an outpatient, single-center, open-label, flexible dose-escalation study design.

DETAILED DESCRIPTION:
This dose-escalation study will examine HLD100 in 24 subjects.

The subjects (n=24) will be tested with HLD100 in ascending doses from 10mg up to 40mg.

This study will be divided into several phases: Screening, Active Treatment and Follow-Up. All visits have a 2 day window to allow for scheduling.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of ADHD as defined by DSM-5 criteria with confirmation using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
* Subjects must demonstrate mild-to-moderate impairment of ADHD symptoms and function per the following at screening (V1) and/or baseline (V2):

  * ADHD-RS-IV score at or above the 90th percentile normalized for sex and age in total score and ≥24 at Baseline;
  * CGI-S score ≥4;
* Subject body weight must be ≥20 kg.
* Subject must be considered clinically appropriate for treatment with amphetamine and HLD100, including prior treatment experience with an amphetamine product, and ability to swallow treatment capsules.

Exclusion Criteria:

* History of, or current, medical condition or laboratory result which, in the opinion of the investigator, unfavorably alters the risk-benefit of study participation, may jeopardize subject safety, or may interfere with the satisfactory completion of the study and study-related procedures.
* Serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, or other cardiac problems that may place the subject at increased vulnerability to the sympathomimetic effects of a stimulant drug.
* History of seizure disorder (except febrile seizures prior to age 5 and with last occurrence at least 1 year prior to study participation), Tourette's disorder, or intellectual disability of minor severity or greater (DSM-5 criteria).
* History of psychosis, bipolar disorder, anorexia nervosa, bulimia, or suicide attempt. Current depression, anxiety, conduct/behavior disorder, substance use disorder, or other psychiatric condition which, in the investigator's opinion, may jeopardize subject safety or may interfere with the satisfactory completion of the study and study-related procedures.
* Active suicidal ideation as evidenced by an ideation score of 2 or greater on the C-SSRS.
* History of severe allergic reaction or intolerance to amphetamine.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-12-18 (Actual); Study Completion 2016-12-27 (Actual)

PRIMARY OUTCOMES:
Dose Escalation to determine optimal dosage for clinical effects | 6 weeks
  Primary outcome is the determination of the dose achieving optimal clinical effect in a safe and tolerable manner

SECONDARY OUTCOMES:
Safety (AEs, ECG, laboratory parameters, physical examinations) | 48 hours
  Safety endpoints include treatment-emergent adverse events (TEAEs), vital signs, electrocardiogram (ECG) parameters, physical examination, and the C-SSRS.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Center for Psychiatry & Behavoural Medicine
Locations (1):
- Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No